CLINICAL TRIAL: NCT04550143
Title: Diaphragm Dysfunction and Peripheral Muscle Wasting in Septic Shock Patients: Exploring Their Relationship Over Time Using Ultrasound Technology
Brief Title: Muscle Ultrasound Study in Shock Patients
Acronym: MUSiShock
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Karim Bendjelid, Professor, University Hospital, Geneva
Other Study IDs: 2020-00452
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Septic Shock
Keywords: Muscle ultrasound; Intensive care unit-acquired weakness; Diaphragm dysfunction; Mechanical ventilation; Weaning; Sepsis; Critical illness
MeSH Terms: conditions — Shock, Septic; Sepsis; Critical Illness | interventions — antigens, CD200

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Septic Shock
  Interventions: Other: Diaphragm ultrasound (DUS); Other: Peripheral Muscle Ultrasound (PMUS); Other: Airway occlusion pressure (P0.1); Other: Medical Research Council (MRC) sum score

INTERVENTIONS:
Other: Diaphragm ultrasound (DUS) — DUS assessments of diaphragmatic thickness (TDI), thickness fraction (TFDI) and shear modulus (SMDI), this last measured by shear-wave elastography (SWE), will be performed for both right and left hemi-diaphragms.
  A landmark between the 8th and 10th intercostal space in the mid-axillary or antero-axillary line, 0.5-2 cm below the costophrenic sinus, will be used. Here, the diaphragm can be seen as the less echogenic structure between two echogenic lines; TDI (cm) will be the calculated as the distance between the two lines at the end of expiration and TFDI as the rate of change between end-expiration and end-inspiration thicknesses (TFDI = "thickness at end inspiration" - "thickness at end-expiration" / "thickness at end-expiration", %).
  SMDI will assess muscle's stiffness. For each image, a region of interest covering the widest possible surface of diaphragm and allowing an acquisition frequency of 2Hz will be set; results will be retrieved in kilopascals (kPa).
  Other Names: Diaphragm ultrasonography
Other: Peripheral Muscle Ultrasound (PMUS) — PMUS assessments of quadriceps rectus femoris (RF) muscle cross-sectional area (CSARF), echogenicity (ECHORF) and shear modulus (SMRF), this last measured by shear-wave elastography (SWE), will be performed.
  Probe will be placed perpendicularly to the anterior plane of the thigh, in 2 anatomical points, as follows:
  (i) in the midpoint between the anterior superior iliac spine and the upper pole of the patella and (ii) the border of the lower 1/3 and upper 2/3 between the anterior superior iliac spine and the upper pole of the patella.
  CSARF (cm2) will be calculated by outlining the area under the muscle hyperechoic line (aponeurosis). For ECHORF (differences in grey-scale images), the analysis of a region of interest (ROI) of 2cm x 2cm will be performed.
  For SMRF (kPa), a ROI covering the widest possible area of the RF and allowing an acquisition frequency of 2Hz will be set for analysis.
  All assessments will be performed with minimal compression and a copious amount of water-gel.
  Other Names: Muscle ultrasonography
Other: Airway occlusion pressure (P0.1) — P0.1 is "the pressure developed in the occluded airway 100 milliseconds after the onset of inspiration". Its use doesn't require any additional equipment since it can be easy measured by using patient's ventilator.
  For the measurement itself, patients will be in semi-recumbent position (head elevation between 30° and 45°) with knee extended in neutral position and will be asked to stay as relaxed as possible. After 5 minutes breathing without any interruption or disturbance, 4 measurements will be observed and recorded as displayed on the ventilator screen.
Other: Medical Research Council (MRC) sum score — This is a manual muscle strength testing tool, used very often in the ICU setting. It's based on the assessment of the following muscle groups: shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and dorsiflexion of the ankle, all scored bilaterally. Muscle strength is graded as follows: 0, "no visible/palpable contraction"; 1, "visible/palpable contraction without movement of the limb"; 2, "movement of the limb, but not against gravity"; 3, "movement against gravity"; 4, "movement against gravity and some resistance"; 5, "normal".
  The sum score ranges between 0 and 60 (between 0 and 5, in 12 muscle groups), with a score <48 indicating the presence of weakness.
  Other Names: MRC muscle strength score

SUMMARY:
Intensive Care Unit (ICU) patients are known to lose muscle mass and function for many reasons, ranging from prolonged immobilization, to the effects of ICU treatments such as mechanical ventilation (MV), to the critical illness itself. Ultrasonography (US) is widely used in the ICU setting and has greatly evolved in the last decades, since it allows the non-invasive assessment of different structures, using radiation-free and user-friendly technology; its application for the assessment or the skeletal muscle is a promising tool and might help detecting muscle changes and thus several dysfunctions during early stages of ICU stay.

By using skeletal muscle ultrasound at both diaphragm and peripheral levels, the overall aim of this study is to improve knowledge in the early detection of muscle dysfunction and weakness , and their relationship with mechanical ventilation weaning and muscle strength, in critically ill patients suffering from septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (> 18 years old) admitted to the ICU
2. with a diagnosis of septic shock
3. a SOFA score equal or superior to 8 points, at ICU admission
4. blood lactate concentration above 2 mmol/L, at ICU admission
5. expected to have more than 48h of mechanical ventilation (estimated by the attending physician)
6. expected to stay more than 5 days in the unit (estimated by the attending physician)
7. able to walk prior to ICU admission / walking aids accepted;

Exclusion Criteria:

1. pregnancy
2. lower limb amputation, fixators or open wounds
3. thoracic fixators or open wounds
4. diagnosed neuromuscular or central nervous system diseases
5. being transferred from another ICU
6. spinal cord injury
7. diaphragm pacemaker
8. palliative goals of care
9. cancers derived sarcopenia
10. cachexia
11. anorexic disorders (protein-energy malnutrition)
12. intellectual or cognitive impairments, limiting the ability to follow instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research project will include any adult patient (> 18 years old) admitted to the ICU (University Hospitals of Geneva, HUG) with a diagnosis of septic shock, respecting the pre-defined inclusion and exclusion criteria. No restrictions will be applied to the source of infection.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Association between SWE assessment and other muscle ultrasound markers. | Baseline (at 24 hours after ICU admission)
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Association between SWE assessment and other muscle ultrasound markers. | Day 2, after ICU admission
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Association between SWE assessment and other muscle ultrasound markers. | Day 3, after ICU admission
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Association between SWE assessment and other muscle ultrasound markers. | Day 4, after ICU admission
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Association between SWE assessment and other muscle ultrasound markers. | Day 5, after ICU admission
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Association between SWE assessment and other muscle ultrasound markers. | Extubation day, approximately 7 days
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Association between SWE assessment and other muscle ultrasound markers. | Weekly (1x/week), counting from day 6 of ICU stay until ICU discharge (approximately 10 days)
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Association between SWE assessment and other muscle ultrasound markers. | ICU discharge, approximately 10 days
  To explore the existence of an association between SWE assessment and other muscle ultrasound markers (TDI, TFDI, CSARF and ECHORF) for each muscle (diaphragm and quadriceps rectus femoris muscles) over the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.

SECONDARY OUTCOMES:
Association between the rate change (%) in DUS and PMUS assessments. | Time-points of assessment relating to baseline (ICU admission) values.
  The association between the rate change (%) in DUS (TDI, TFDI and SMDI) and PMUS (CSARF, ECHORF and SMRF) markers over time, during the ICU stay, in adult patients (> 18 years old) admitted for a septic shock.
Weaning success/failure predictive model. | Between ICU admission and extubation moment.
  The analysis of a combined model comprising, among other ICU variables, one DUS marker (TDI, TFDI and SMDI) and one PMUS marker (CSARF, ECHORF and SMRF) to predict weaning success/failure, in adult patients (> 18 years old) admitted to the ICU for a septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Bendjelid, MD, PhD, Principal Investigator — Hôpitaux Universitaires de Genève (HUG) / Université de Genève (UNIGE)
Locations (1):
- Service de Soins Intensifs, Hôpitaux Universitaires de Genève (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Puthucheary ZA, Phadke R, Rawal J, McPhail MJ, Sidhu PS, Rowlerson A, Moxham J, Harridge S, Hart N, Montgomery HE. Qualitative Ultrasound in Acute Critical Illness Muscle Wasting. Crit Care Med. 2015 Aug;43(8):1603-11. doi: 10.1097/CCM.0000000000001016. PMID 25882765
- [Background] Dres M, Dube BP, Mayaux J, Delemazure J, Reuter D, Brochard L, Similowski T, Demoule A. Coexistence and Impact of Limb Muscle and Diaphragm Weakness at Time of Liberation from Mechanical Ventilation in Medical Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Jan 1;195(1):57-66. doi: 10.1164/rccm.201602-0367OC. PMID 27310484
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Bachasson D, Dres M, Nierat MC, Gennisson JL, Hogrel JY, Doorduin J, Similowski T. Diaphragm shear modulus reflects transdiaphragmatic pressure during isovolumetric inspiratory efforts and ventilation against inspiratory loading. J Appl Physiol (1985). 2019 Mar 1;126(3):699-707. doi: 10.1152/japplphysiol.01060.2018. Epub 2019 Feb 7. PMID 30730816
- [Background] Flatres A, Aarab Y, Nougaret S, Garnier F, Larcher R, Amalric M, Klouche K, Etienne P, Subra G, Jaber S, Molinari N, Matecki S, Jung B. Real-time shear wave ultrasound elastography: a new tool for the evaluation of diaphragm and limb muscle stiffness in critically ill patients. Crit Care. 2020 Feb 3;24(1):34. doi: 10.1186/s13054-020-2745-6. PMID 32014005
- [Background] Quenot JP, Binquet C, Kara F, Martinet O, Ganster F, Navellou JC, Castelain V, Barraud D, Cousson J, Louis G, Perez P, Kuteifan K, Noirot A, Badie J, Mezher C, Lessire H, Pavon A. The epidemiology of septic shock in French intensive care units: the prospective multicenter cohort EPISS study. Crit Care. 2013 Apr 25;17(2):R65. doi: 10.1186/cc12598. PMID 23561510
- [Background] SepNet Critical Care Trials Group. Incidence of severe sepsis and septic shock in German intensive care units: the prospective, multicentre INSEP study. Intensive Care Med. 2016 Dec;42(12):1980-1989. doi: 10.1007/s00134-016-4504-3. Epub 2016 Sep 29. PMID 27686355
- [Derived] Neto Silva I, Duarte JA, Perret A, Dousse N, Wozniak H, Bollen Pinto B, Giraud R, Bendjelid K. Diaphragm dysfunction and peripheral muscle wasting in septic shock patients: Exploring their relationship over time using ultrasound technology (the MUSiShock protocol). PLoS One. 2022 Mar 28;17(3):e0266174. doi: 10.1371/journal.pone.0266174. eCollection 2022. PMID 35344570